CLINICAL TRIAL: NCT03202303
Title: Cannabidivarin (CBDV) vs. Placebo in Children With Autism Spectrum Disorder (ASD)
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Montefiore Medical Center (Other)
Collaborators: United States Department of Defense (U.S. Federal Agency); GW Pharmaceuticals Ltd (Industry); Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2017-8538; AR160104 (Other Grant/Funding Number: Department of Defense (DOD)); G32379 (Other Grant/Funding Number: GW Pharmaceuticals)
Record Dates: First submitted 2017-06-27; First posted 2017-06-28 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-10

CONDITIONS: Autism Spectrum Disorder
Keywords: Autism; Irritability; Cannabinoids
MeSH Terms: conditions — Autism Spectrum Disorder; Autistic Disorder | interventions — cannabidivarin

STUDY DESIGN:
Intervention Model Description: Phase 2, 12-week double-blind, randomized, placebo-controlled trial
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Double-Blind
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Cannabidivarin (CBDV) (Experimental): Weight-based dosing of 10 mg/kg/day of CBDV for 12 weeks
  Interventions: Drug: Cannabidivarin
- Matched Placebo (Placebo Comparator): Weight-based dosing of 10 mg/kg/day of placebo for 12 weeks
  Interventions: Drug: Matched Placebo

INTERVENTIONS:
Drug: Cannabidivarin — Weight-based dosing of 10 mg/kg/day of CBDV
  Other Names: CBDV
  Arms: Cannabidivarin (CBDV)
Drug: Matched Placebo — Weight-based dosing of 10 mg/kg/day of placebo
  Other Names: Placebo
  Arms: Matched Placebo

SUMMARY:
This trial aims to study the efficacy and safety of cannabidivarin (CBDV) in children with ASD.

DETAILED DESCRIPTION:
There is a clear unmet need for new therapeutics to treat irritability in children with ASD that do not have the metabolic and weight adverse event profiles of the currently approved treatments. Cannabidivarin (CBDV) is a nonpsychoactive phytocannabinoid and a safe variant of Cannabidiol (CBD). It has no appreciable tetrahydrocannabinol (THC) [less than 0.01%], has been shown to have no impact on weight or metabolism, and improves both social and cognitive functioning in animal models of idiopathic and syndromal autism (Fragile X, Rett Syndrome, Angelman Syndrome). The CDC currently estimates 1 in 59 children have ASD. ASD is characterized by deficits in social communication, irritability, repetitive behaviors, impulsivity, temper tantrums, and high caregiver burden. Currently, the only FDA-approved medications for symptoms of ASD are aripiprazole and risperidone, both of which are indicated for irritability in pediatric ASD. These medications are effective but are associated with considerable side effects with long term treatment in this chronic developmental disorder, including weight gain, metabolic syndrome and the risk of type 2 diabetes, prolactin elevation and growth of breast tissue, extrapyramidal symptoms and the risk of tardive dyskinesia. The anticonvulsant divalproex sodium (valproate/VPA) also significantly reduces irritability and repetitive behaviors in individuals with ASD. Although VPA is efficacious for pediatric epilepsy and some symptoms of ASD, it also has significant side effects, including weight gain, sedation and nausea. CBDV, like VPA, is effective in the treatment of pediatric epilepsy, and ASD mouse models demonstrate potential mechanisms for treatment with CBDV, including potential therapeutic effects on repetitive behaviors, irritability, sociability, and quality of life, and the capacity to reduce inflammation. This study aims to examine the efficacy and safety of cannabidivarin (CBDV) with a primary aim of studying its effect on irritability in children with ASD.

STUDY DESIGN: This is a 12-week randomized, double-blind study of CBDV vs. placebo in 100 child and adolescent subjects aged 5 to 18 years with a diagnosis of ASD.

ELIGIBILITY:
Inclusion Criteria

1. Male or Female pediatric outpatients aged between and including ages 5 to 18. Diagnosis of Autism Spectrum Disorder (ASD) confirmed by the ADOS-2 and DSM-5 criteria.*During special circumstances (e.g. COVID-19 pandemic) where the ADOS-2 cannot be performed due to site restrictions (e.g. mandatory use of face masks), eligibility can be confirmed using the Autism Diagnostic Interview, Revised (ADI-R)
2. Aberrant Behavior Checklist (ABC) - Irritability Subscale (ABC-I) score of 18 or greater at screening visit.
3. Social Responsiveness Scale (SRS) score of 66T or higher at screening visit.
4. Clinical Global Impression Scale - Severity (CGI-S) score of 4 or higher at screening.
5. Stable pharmacologic, educational, behavioral and/or dietary interventions for 4 weeks prior to randomization and for the duration of the study.
6. Physical exam and laboratory results that are within normal range for individuals with ASD.
7. Presence of a parent/caregiver/guardian that is able to consent for their participation and complete assessments regarding the child's development and behavior throughout the study. Child Assent will be obtained if the subject is 7 years of age or older and has the mental capacity to understand and sign a written assent form and/or give verbal assent.

Exclusion Criteria

1. Exposure to any investigational agent in the 30 days prior to randomization.
2. Prior chronic treatment with CBD, CBDV or an endocannabinoid treatment.
3. Positive testing for THC or other drugs of abuse via urine testing at the screening visit or baseline visits upon repeat confirmation testing.
4. Recent history of drug abuse including marijuana/cannabis use in the past 3 months.
5. Diagnosis of a known genetic disorder (ie. Prader-Willi Syndrome, Angelman Syndrome etc.).
6. A primary psychiatric diagnosis other than ASD, including bipolar disorder, psychosis, schizophrenia, Post-Traumatic Stress Disorder (PTSD) or Major Depressive Disorder (MDD). These patients will be excluded due to potential confounding results.
7. A medical condition that severely impacts the subject's ability to participate in the study, interferes with the conduct of the study, confounds interpretation of study results or endangers the subject's well-being.
8. A known diagnosis of Rett Syndrome or Childhood Disintegrative Disorder, or marked sensory impairment such as deafness or blindness.
9. Subjects who have had changes in allied health therapies, behavioral or educational interventions within four weeks prior to randomization other than those associated with school holidays.
10. Subjects who have had changes in medications or medication doses within four weeks of randomization. Renal, pancreatic, or hematologic dysfunction as evidenced by values above upper limits of normal for BUN/creatinine, or values twice the upper limit of normal for serum lipase and amylase, platelets <80,000 /mcL, or WBC<3.0 103 /mcL
11. Liver dysfunction manifested by > 2 X UNL values of AST or ALT
12. ECG abnormality at baseline screening or clinically significant postural drop in systolic blood pressure at screening. If the initial screening ECG show a QTcB of greater than 460 msec, then 2 additional ECGs will be conducted in the same sitting, 5 minutes apart. If not recognized at screening, then a full triplicate repeat showing an average QTcB of 460 msec or less to meet all inclusion/exclusion criteria. Female subjects who are pregnant will be excluded from the study. If a female subject is able to become pregnant, she will be given a serum pregnancy test before entry into the study. Female subjects will be informed not to become pregnant while taking CBDV. Female subjects must tell the investigator and consult an obstetrician or maternal-fetal specialist if they become pregnant during the study.
13. Known allergy to sesame oil

Ages: 5 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-04-12 (Actual); Primary Completion 2027-02 (Estimated); Study Completion 2027-02 (Estimated)

PRIMARY OUTCOMES:
Aberrant Behavior Checklist-Irritability (ABC-I) Subscale | Change from Baseline to Week 12 (Change over 12 weeks)
  Change in aberrant behavior from baseline will be assessed using the irritability subscale of the ABC. The ABC is an informative rating instrument that was empirically derived by principal component analysis to measure behavior in those with developmental disability and autism spectrum disorder (ASD). The ABC-I will be completed by any adult who knows the patient well, such as a parent/caregiver. The ABC-I subscale consists of 15 items that address the presence of aggression, tantrums, and/or self-injury. Scores for each item on the subscale range from 0 (no problem at all) to 3 (problem is severe in degree), yielding an overall possible score for the subscale from 0-45, such that higher scores are indicative of increased severity of irritability. Scores will be summarized by study arm using basic descriptive statistics.

SECONDARY OUTCOMES:
Repetitive Behavior Scale-Revised (RBS-R) | Change in RBS-R from Baseline to Week 12 (Change over 12 weeks)
  Change in repetitive behavior from baseline will be assessed using the RBS-R, a 43-item self-report instrument that is used to measure the breadth of repetitive behaviors specific to autism spectrum disorder (ASD) symptomatology. The 43 items encompass 6 behavioral subscales including: Stereotypic (6 items); Self-injurious (8 items); Compulsive (8 items); Ritualistic (6 items); Sameness (11 items); and Restricted Behavior (4 items). A list of behaviors will be presented and the parent will be asked to choose a score that best describes how much of a problem the behavior has been over the last month. Behaviors are rated on a 4-point scale: 0 (behavior does not occur), 1 (behavior occurs and is a mild problem), 2 (behavior occurs and is a moderate problem) and 3 (behavior occurs and is a severe problem). Higher scores reflect increased severity of repetitive behavior for that scale. Scores for each of the 6 subscales will be summarized by arm using basic descriptive statistics.
Montefiore Einstein Rigidity Scale-Revised (MERS-R) | Change in MERS-R from Baseline to Week 12 (Change over 12 weeks)
  Change in rigidity from baseline will be assessed using the MERS-R. MERS-R is designed to assess three domains of rigid behavior in children (and adults) with ASD: Behavioral Rigidity (e.g., insistence on sameness, things must be done his/her way, etc.); Cognitive Rigidity (e.g., special interests, inflexible adherence to rules, etc.); and Protest (in response to deviation from rigidity; e.g., verbal objection, tantrum, physical aggression). MERS-R is a clinician-rated scale and will only be completed only for subjects who display rigid behaviors at baseline, and study visits during week 4, week 8, and week 12. The MERS-R consists of 43 items. Each item is scored based on a 4-point scale ranging from 0 (no problem) to 3 (severe problem) for rigid behaviors displayed over the past month, yielding an overall MERS-R score of 0-129. Higher scores are associated with more severe rigidity. Scores will be summarized by study arm using basic descriptive statistics.
Aberrant Behavior Checklist-Social Withdrawal (ABC-SW) Subscale | Change in ABC-SW from Baseline to Week 12 (Change over 12 weeks)
  Change in aberrant behavior from baseline will also be evaluated using the Social Withdrawal subscale of the Aberrant Behavior Checklist (ABC). The ABC is an informant rating instrument that measures behavior in individuals with developmental disability and ASD. The ABC-SW scale measures behavior using a 4-point severity scale, ranging from 0-3, where parents rate aberrant behaviors as 0 = no problem at all, 1 = behavior is a problem but in a slight degree, 2 = problem is moderately serious, and 3 = problem is severe in degree, such that higher scores are associated with increased severity of social withdrawal, for an overall possible score of 0-48. Scores will be summarized by study arm using basic descriptive statistics.
Pediatric Quality of Life Inventory (PedsQL) Family Impact Module | Change in PedsQL from Baseline to Week 12 (Change over 12 weeks)
  Change in quality of life is assessed using the PedsQL family impact module, a 36-item self-report caregiver form used to measure caregiver functioning. PedsQL encompasses 6 scales: Physical Functioning (6 items), Emotional Functioning (5 items), Social Functioning (4 items), Cognitive Functioning (5 items), Communication (3 items), Worry (5 items) and 2 scales measuring caregiver-reported family functioning: Daily Activities (3 items) and Family Relationships (5 items). Each item is scored using a 5-point scale ranging from 0 (never a problem) to 4 (always a problem). Items are then reverse-scored and transformed to a 0-100 scale (0 = 100, 1 = 75, 2 = 50, 3 = 25, 4 = 0), such that higher scores indicate better functioning (less negative impact). Scale Scores are computed as the sum of the items divided by the number of items answered (to account for missing data). If >50% of the items in the scale are missing, a scale score is not computed. Scores will be summarized by study arm.
Vineland Adaptive Behavior Scale, Third Edition (VABS-3) | Change in VABS-3 from Baseline to Week 12 (Change over 12 weeks)
  Change in adaptive behavior from baseline will be assessed using the VABS-3. The VABS-3 is an instrument that measures adaptive behavior across 5 domains: communication, daily living skills, socialization, motor skills, and maladaptive behavior of individuals with developmental disabilities. The Survey Interview Form (semi-structured interview) will be administered to a participant's reliable caregiver in this study, during which the interviewer will ask the caregiver open ended questions relating to the subject's activities and behavior. Scoring involves assigning points (0, 1, or 2) to each item based on the responses to the questions. These scores are then compared to normative data to determine the individual's standing relative to peers. Higher scores are generally indicative of better adaptive behavior. Scores will be summarized by study arm using basic descriptive statistics.
Clinical Global Impressions - Improvement (CGI-I) | Change in CGI-I from Baseline to Week 12 (Change over 12 weeks)
  The degree of change of in condition from baseline will be assessed using the CGI-I scale. The CGI-I is a clinician-rated global measure of improvement scale used to assess the degree of symptom change in a patient relative to baseline condition. It consists of a 7-point scale as follows: 1 = very much improved, 2 = much improved, 3 = minimally improved, 4 = no change, 5 = minimally worse, 6 = much worse, and 7 = very much worse, such that lower scores are indicative of increased symptom improvement. Scores will be summarized by study arm using basic descriptive statistics.

CONTACTS AND LOCATIONS:
Overall Officials: Eric Hollander, MD, Principal Investigator — Montefiore Medical Center/Albert Einstein College of Medicine
Locations (2):
- United States (2):
  - New York University (NYU) Langone, New York, New York
  - Montefiore Medical Center, The Bronx, New York

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Ferretti CJ, Cook BL, Mahant AM, Chu P, Zhao Y, Taylor BP, Herold BC, Hollander E. Cognitive inflexibility and immunome biomarkers in children with autism spectrum disorder. Neurosci Appl. 2024 May 4;3:104071. doi: 10.1016/j.nsa.2024.104071. eCollection 2024. PMID 40656115